CLINICAL TRIAL: NCT04828044
Title: Microwave Ablation of Breast Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Lack of sufficient funding
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Other Study IDs: 12-028 MWA - Breast Tumors
Record Dates: First submitted 2012-09-12; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tumors
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimens will be evaluated and stored as standard surgical pathology specimens by the St. Joseph Hospital Department of Pathology. Additional tissue needed for tumor marker studies will be obtained prior to MWA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Microwave Ablation/ Coagulation Arm: These patients will receive microwave ablation using MedWaves Microwave Ablation/ Coagulation System.
  Interventions: Device: Microwave Ablation/ Coagulation Arm

INTERVENTIONS:
Device: Microwave Ablation/ Coagulation Arm — An 11-gauge microwave probe from MedWaves, Inc., will be placed in the tumor. An ablation lesion will then be generated at the appropriate power (10-35 watts) to maintain up to 130C degrees at the MW applicator tip thermocouple for 10 minutes duration. Palpation and/or ultrasound may be used to place the MWA needle and monitor the progress of the microwave ablation.
  Other Names: Medwaves Microwave Ablation/ Coagulation System

SUMMARY:
The purpose of this protocol is to pathologically evaluate the amount of destruction of cancer cells by Microwave Ablation (MWA) in primary breast tumors.

DETAILED DESCRIPTION:
Minimally invasive surgical alternatives are becoming more attractive for the treatment of malignancy due to improvements in technology, reduced costs and reduced morbidity. The main objective of this protocol is to determine the extent of ablation based on time and power parameters of the MedWaves in breast cancers. This would be accomplished in patients diagnosed with breast cancer who are already scheduled for breast cancer surgery. Prior to the surgical removal of the cancer, the microwave antenna would be inserted into the tumor under ultrasound guidance (either percutaneously or open). The tumor would be ablated, and then surgically resected in a standard, curative fashion.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of primary breast tumor for which a surgical resection (excisional, biopsy, segmentectomy or mastectomy) is planned.
* Tumor is palpable or visible on ultrasound or both
* All participants need to be fully able to give informed consent

Exclusion Criteria:

* Gender: male
* Mental or legal incompetence
* Impaired decision-making capacity
* Pregnant women may not participate
* Implanted Pacemaker

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of primary breast tumor for which a surgical resection (excisional, biopsy, segmentectomy or mastectomy) is planned.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Amount of tissue destruction with MedWaves Microwave Ablation/ Coagulation System. | 30 days
  Measure tissue destruction with the MedWaves Microwave Ablation/ Coagulation System through pathological review of destruction.

SECONDARY OUTCOMES:
Provide the differences between percutaneous and open Microwave Ablation | 30 Days
  Evaluate differences between percutaneous and open Microwave Ablation through pathological review and patient follow-up.
Amount of toxicity of microwave ablation in patients. | 30 Days
  Measure toxicity of Microwave Ablation through patient follow-up and assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Wagman, M.D., Principal Investigator — St. Joseph Hospital of Orange
Locations (1):
- St. Joseph Hospital of Orange, Orange, California, United States